CLINICAL TRIAL: NCT05770895
Title: A Phase 1a/1b Study to Evaluate the Safety and Tolerability of Repeated Doses of Nonreplicating Arenavirus Vector Therapeutic Vaccines GS-2829 and GS-6779 in Healthy Participants and Participants With Chronic Hepatitis B (CHB)
Brief Title: Study of HBV Therapeutic Vaccines GS-2829 and GS-6779 in Healthy Participants and Participants With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-642-5670
Record Dates: First submitted 2023-03-01; First posted 2023-03-16 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 injections) (Experimental): Healthy participants will receive a single low dose of GS-2829 (≥ 0.5 x 10^6 focus-forming unit (FFU)/mL) or placebo as intramuscular (IM) injection on Days 1 and 57.
  Interventions: Biological: GS-2829; Biological: Placebo
- Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 injections) (Experimental): Healthy participants will receive a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL) or placebo as IM injection on Days 1 and 57.
  Interventions: Biological: GS-6779; Biological: Placebo
- Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 cycles) (Experimental): Healthy participants will receive a single low dose of GS-2829 (≥ 0.5 x 10^6 FFU/mL) or placebo as IM injection on Days 1 and 57; and a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL) or placebo as IM injection, on Days 29 and 85.
  Interventions: Biological: GS-2829; Biological: GS-6779; Biological: Placebo
- Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 cycles) (Experimental): Healthy participants will receive a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection, on Days 1 and 57; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection, on Days 29 and 85.
  Interventions: Biological: GS-2829; Biological: GS-6779; Biological: Placebo
- Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 cycles) (Experimental): Healthy participants will receive a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection on Days 1, 57 and 113; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection on Days 29, 85 and 141.
  Interventions: Biological: GS-2829; Biological: GS-6779; Biological: Placebo
- Phase 1b : Cohort 5 (VS Participants with CHB) : GS-2829 and GS-6779 Low Dose (2 cycles) (Experimental): Virally suppressed (VS) participants with Chronic Hepatitis B (CHB) will receive a single low dose of GS-2829 (≥ 0.5 x 10^6 FFU/mL) or placebo as IM injection on Days 1 and 57; and a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL) or placebo as IM injection on Days 29 and 85.
  Interventions: Biological: GS-2829; Biological: GS-6779; Biological: Placebo
- Phase 1b : Cohort 6 (VS Participants with CHB) : GS-2829 and GS-6779 High Dose (2 cycles) (Experimental): VS participants with CHB will receive a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection on Days 1 and 57; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection on Days 29 and 85.
  Interventions: Biological: GS-2829; Biological: GS-6779; Biological: Placebo
- Phase 1b : Cohort 7 (VS Participants with CHB) : GS-2829 and GS-6779 High Dose (3 cycles) (Experimental): VS participants with CHB will receive a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection on Days 1, 57 and 113; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) or placebo as IM injection on Days 29, 85 and 141.
  Interventions: Biological: GS-2829; Biological: GS-6779; Biological: Placebo

INTERVENTIONS:
Biological: GS-2829 — Administered intramuscularly
  Arms: Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 injections); Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 cycles); Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 cycles); Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 cycles); Phase 1b : Cohort 5 (VS Participants with CHB) : GS-2829 and GS-6779 Low Dose (2 cycles); Phase 1b : Cohort 6 (VS Participants with CHB) : GS-2829 and GS-6779 High Dose (2 cycles); Phase 1b : Cohort 7 (VS Participants with CHB) : GS-2829 and GS-6779 High Dose (3 cycles)
Biological: GS-6779 — Administered intramuscularly
  Arms: Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 injections); Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 cycles); Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 cycles); Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 cycles); Phase 1b : Cohort 5 (VS Participants with CHB) : GS-2829 and GS-6779 Low Dose (2 cycles); Phase 1b : Cohort 6 (VS Participants with CHB) : GS-2829 and GS-6779 High Dose (2 cycles); Phase 1b : Cohort 7 (VS Participants with CHB) : GS-2829 and GS-6779 High Dose (3 cycles)
Biological: Placebo — Administered intramuscularly

SUMMARY:
The goal of this clinical study is to learn more about GS-2829 and GS-6779 in healthy participants and participants with CHB.

ELIGIBILITY:
Key Inclusion Criteria:

Phase 1a and 1b:

* Body mass index (BMI) of ≤ 32.0 kg/m^2.
* Non-diabetic without impaired glucose tolerance.
* No evidence of cardiac disease based on 12 lead electrocardiogram (ECG).

Phase 1a (Healthy Individuals) only:

* Aged 18 through 60 years.
* No prior history of Hepatitis B infection with a negative hepatitis B surface antigen (HBsAg) and Hepatitis B (HBV) core antibody.

Phase 1b (Virally Suppressed chronic hepatitis B (CHB) Individuals)):

* Aged 18 through 65 years.
* Documented CHB and HBsAg ≤ 5000 IU/mL at screening.
* No evidence of advanced fibrosis by Fibroscan (defined as Fibroscan < 9 kilo pascal (kPa) within 6 months of screening).
* Diagnosed with CHB on suppressive oral antiviral for ≥ 6 months.
* Must have received an approved HBV-active oral antiviral agent for ≥ 6 months prior to screening with HBV DNA below lower limit of quantification (LLOQ) for ≥ 3 months prior to screening and with no plan to stop HBV-active antivirals during the study.

Key Exclusion Criteria:

Phase 1a and 1b:

* Use of any systemic antibiotics within 30 days of screening.
* Receipt of any HBV vaccine within 12 months of screening visit or planning HBV vaccination during the study period.
* Receipt of any investigational product within 3 months or vaccine within 3 months of screening (with the exception of influenza and severe acute respiratory syndrome (SARs) coronavirus (COV) - 2 (SARS-CoV-2) vaccines, which if needed, should be administered at least 14 days before or after an investigational product administration).
* Receipt of immunoglobulin or other blood products within 3 months of screening.
* Positive serum pregnancy test at screening or positive urine pregnancy on Day 1.
* Have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to screening or is expected to receive these agents during the study (eg, corticosteroids, immunoglobulins, other immune or cytokine-based therapies).
* Participation in any other clinical study (including observational studies) without prior approval from the sponsor is prohibited while participating in the study.

Note - Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- New Zealand Clinical Research (NZCR), Auckland, New Zealand
- Taiwan (8):
  - Chia-Yi Christian Hospital, Chiayi City
  - St. Martin De Porres Hospital, Chiayi City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gane E J et al. Safety, tolerability and immunogenicity of GS-2829 and GS-6779, a novel arenaviral vectored therapeutic hepatitis B vaccine: results from a phase 1a study in healthy participants. Poster THU-246. Presented at European Association for the Study of the Liver (EASL), 07-10 May 2025, Amsterdam, The Netherlands. J Hepatol 2025;82(S1):S831.
- [Background] Gane E J, et al. Safety, tolerability, immunogenicity, and antiviral efficacy of GS-2829 and GS-6779, a novel, arenaviral-vectored, therapeutic hepatitis B vaccine: Results from a phase 1b study in virally suppressed patients with chronic hepatitis B. *Hepatology*. 2025;72(Suppl 1):197. Presented at: AASLD The Liver Meeting; November 7-11, 2025; San Diego, CA.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-642-5670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in New Zealand and Taiwan.
Pre-assignment Details: 148 participants (114 in Phase 1a and 34 in Phase 1b) were screened.
Groups:
- Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections): Healthy participants received a single low dose of GS-2829 (≥ 0.5 x 10^6 FFU/mL) as Intramuscular (IM) injection on Days 1 and 57.
- Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections): Healthy participants received a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL) as IM injection on Days 1 and 57.
- Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles): Healthy participants received a single low dose of GS-2829 (≥ 0.5 x 10^6 FFU/mL) as IM injection on Days 1 and 57; and a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL) as IM injection on Days 29 and 85.
- Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles): Healthy participants received a single high dose of GS-2829 (0.5 mL of a undiluted ≥ 0.5 x 10^7 FFU/mL) as IM injection on Day 1 and Day 57; and single high dose of GS-6779 (0.5 ml of a undiluted ≥ 0.5 x 10^7 FFU/mL) as IM injection on Day 29 and Day 85.
- Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles): Healthy participants received a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) as IM injection on Days 1, 57 and 113; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) as IM injection on Days 29, 85 and 141.
- Phase 1a: Placebo : Healthy Participants: Healthy participants who received placebo pooled across Phase 1 a Cohorts 1-4 and 8 (2 participants per cohort were randomized to placebo).
- Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles): VS participants with CHB received a single low dose of GS-2829 (≥ 0.5 x 10^6 FFU/mL) as IM injection on Days 1 and 57; and a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL ) as IM injection on Days 29 and 85.
- Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles): VS participants with CHB received a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) as IM injection on Days 1 and 57; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) as IM injection on Days 29 and 85.
- Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles): VS participants with CHB received a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) as IM injection on Days 1, 57 and 113; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) as IM injection on Days 29, 85 and 141.
- Phase 1b: Placebo : VS CHB Participants: VS CHB participants who received placebo pooled across Phase 1b Cohorts 5-7 (2 participants per cohort were randomized to placebo).
Period: Overall Study
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants
Started | 8 | 8 | 10 | 8 | 9 | 10 | 8 | 8 | 8 | 6
Completed | 8 | 8 | 8 | 8 | 7 | 10 | 8 | 8 | 8 | 6
Not Completed | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but never treated | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections): Healthy participants received a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL)] as IM injection on Days 1 and 57.
- Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles): Healthy participants received a single low dose of GS-2829 (≥ 0.5 x 10^6 FFU/mL) as IM injection on Days 1 and 57; and a single low dose of GS-6779 (≥ 0.5 x 10^6 FFU/mL) as IM injection, on Days 29 and 85.
- Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles): Healthy participants received a single high dose of GS-2829 (≥ 0.5 x 10^7 FFU/mL) as IM injection, on Days 1 and 57; and a single high dose of GS-6779 (≥ 0.5 x 10^7 FFU/mL) as IM injection, on Days 29 and 85.
- Total: Total of all reporting groups
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 10 | 8 | 8 | 8 | 6 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 9 | 10 | 8 | 8 | 8 | 6 | 81
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.7) | 30 (5.4) | 35 (13.0) | 34 (9.8) | 31 (8.8) | 38 (11.4) | 55 (6.1) | 46 (8.9) | 48 (9.8) | 49 (9.6) | 40 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 7 | 3 | 4 | 3 | 3 | 1 | 4 | 37
  Male | 3 | 6 | 3 | 1 | 6 | 6 | 5 | 5 | 7 | 2 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Not Hispanic or Latino | 7 | 6 | 7 | 5 | 9 | 10 | 8 | 8 | 8 | 6 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 3 | 4 | 4 | 1 | 4 | 8 | 8 | 8 | 6 | 48
  Race: White | 5 | 3 | 3 | 1 | 5 | 4 | 0 | 0 | 0 | 0 | 21
  Race: Other or More Than One Race | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 9
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 8 | 8 | 8 | 8 | 9 | 10 | 3 | 0 | 2 | 1 | 57
  Taiwan | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 6 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as any AE with a start date on or after the study drug start date; or any AE that led to premature discontinuation of study drug. An SAE is defined as an event that, at any dose, results in the following: Death, a life-threatening situation, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or a medically important event or reaction.
Time Frame: First dose date to end of study (followed up to 24 weeks post last dose (up to Day 225 [cohorts 1, 2], Day 253 [cohorts 3, 4, 5, 6], and Day 309 [cohorts 7 and 8])
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 10 | 8 | 8 | 8 | 6
percentage of participants
  Any TEAE | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 90.0 | 75.0 | 62.5 | 75.0 | 50.0
  SAE | 0 | 0 | 0 | 0 | 11.1 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any time postbaseline. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed postbaseline will be considered treatment emergent.
Time Frame: as for outcome 1
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 9 | 10 | 8 | 8 | 8 | 6
percentage of participants | 100.0 | 87.5 | 100.0 | 100.0 | 88.9 | 90.0 | 87.5 | 100.0 | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants With ≥ 3-Fold Increase in Vaccine-Induced Hepatitis B Virus (HBV) Specific T-Cell Responses
Description: Vaccine-induced HBV-specific T cell responses were measured using an interferon-gamma (IFN-γ), enzyme-linked immunospot (ELISpot) assay with a readout of spot forming cells (SFCs) /10^6 peripheral blood mononuclear cells (PBMCs). Total response was the sum of the dimethylsulfoxide (DMSO) -adjusted averages for the 4 HBV peptides (HBV core + HBV polymerase (pol) A + HBV pol B + HBV surface antigen (sAg)). Response was defined as a ≥ 3-fold increase over baseline in vaccine-induced HBV-specific total T cell response (measured using the IFN-γ ELISpot assay). A participant's highest fold-increase postbaseline was utilized for analysis of responder/non-responder. Participants with missing values for fold change over baseline were counted as failures (missing = failure).
Time Frame: Up to 24 weeks post last dose (up to Day 225 [cohorts 1, 2]) or up to 12 weeks post last dose (up to Day 169 [cohorts 3, 4, 5, 6]; Day 225 [cohorts 7 and 8])
Population: Participants in the Immunogenicity Analysis Set were analyzed. The Immunogenicity Analysis Set included all randomized participants who received at least 1 dose of study drug and have at least 1 value for HBV-specific T-cell total response using the interferon gamma (IFN-γ) enzyme-linked immunospot (EliSpot) assay after administration of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 6
percentage of participants | 12.5 | 0.0 | 87.5 | 87.5 | 100.0 | 0.0 | 25.0 | 0.0 | 37.5 | 16.7

4. Secondary Outcome: Mean Peak Levels of Vaccine-Induced HBV Specific T-Cell Responses
Description: Vaccine-induced HBV-specific T cell responses were measured using an IFN-γ ELISpot assay with a readout of SFCs/10^6 PBMCs. Total response was the sum of the DMSO-adjusted averages for the 4 HBV peptides (HBV Core + HBV Pol A + HBV Pol B + HBV sAg). Peak values were the highest posttreatment value for an individual participant and then means were calculated across the participants in a cohort.
Time Frame: as for outcome 3
Population: Participants in the Immunogenicity Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: SFC/10^6 PBMCs
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 6
SFC/10^6 PBMCs | 1154.0 (2427.31) | 196.0 (0.00) | 1677.1 (1748.80) | 2853.7 (2273.66) | 3865.2 (2686.77) | 283.6 (127.68) | 674.4 (411.83) | 401.1 (98.49) | 546.8 (227.56) | 374.7 (258.29)

ADVERSE EVENTS:
Time Frame: Up to Day 225 for Cohorts 1, 2; Up to Day 253 for Cohorts 3, 4, 5, 6; Up to Day 309 for Cohorts 7 and 8
Description: All cause mortality analyzed for All Randomized Analysis Set (participants randomized into study).
  AEs analyzed for Safety Analysis Set (all participants who received at least 1 dose of study drug).
Arm/Group | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1a: Placebo : Healthy Participants | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) | Phase 1b: Placebo : VS CHB Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/8 | 0/9 | 0/10 | 0/8 | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 1/9 | 0/10 | 0/8 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 8/8 | 9/9 | 9/10 | 6/8 | 5/8 | 6/8 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) (N=8) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) (N=8) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) (N=8) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) (N=8) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) (N=9) | Phase 1a: Placebo : Healthy Participants (N=10) | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) (N=8) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) (N=8) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) (N=8) | Phase 1b: Placebo : VS CHB Participants (N=6)
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a : Cohort 1 (Healthy Participants) : GS-2829 Low Dose (2 Injections) (N=8) | Phase 1a : Cohort 2 (Healthy Participants) : GS-6779 Low Dose (2 Injections) (N=8) | Phase 1a : Cohort 3 (Healthy Participants) : GS-2829 and GS-6779 Low Dose (2 Cycles) (N=8) | Phase 1a : Cohort 4 (Healthy Participants) : GS-2829 and GS-6779 High Dose (2 Cycles) (N=8) | Phase 1a : Cohort 8 (Healthy Participants) : GS-2829 and GS-6779 High Dose (3 Cycles) (N=9) | Phase 1a: Placebo : Healthy Participants (N=10) | Phase 1b : Cohort 5 (VS Participants With CHB) : GS-2829 and GS-6779 Low Dose (2 Cycles) (N=8) | Phase 1b : Cohort 6 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (2 Cycles) (N=8) | Phase 1b : Cohort 7 (VS Participants With CHB) : GS-2829 and GS-6779 High Dose (3 Cycles) (N=8) | Phase 1b: Placebo : VS CHB Participants (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival cyst (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 5 | 3 | 6 | 4 | 3 | 3 | 3 | 3 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 2 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0
Injection site discomfort (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 2 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
Injection site induration (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 5 | 5 | 8 | 4 | 3 | 3 | 3 | 2 | 2
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 2 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 6 | 5 | 1 | 1 | 1 | 3 | 1
Medical device pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2 | 4 | 2 | 2 | 0 | 1 | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 5 | 3 | 0 | 2 | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 1 | 7 | 4 | 4 | 2 | 1 | 1 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT05770895/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT05770895/SAP_001.pdf